CLINICAL TRIAL: NCT06588192
Title: Renal Survival in Patients with Lupus Nephritis in Assiut University Hospital: a Single-center Study
Brief Title: Renal Survival in Patients with Lupus Nephritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Soudy Ahmed Hmad, Assistant Lecturer, Assiut University
Other Study IDs: survival in lupus nephritis
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lupus Nephritis (LN)
Keywords: lupus; nephritis
MeSH Terms: conditions — Lupus Nephritis; Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Systemic lupus erythematous is a chronic multifactorial autoimmune disease that affects many organs including kidney. Lupus nephritis is a common manifestation characterized by heterogeneous clinical and histopathological finding and often associate with poor progression and despite potent anti-inflammatory and immunosuppressive therapies still end in CKD or ESRD for too many patient. lupus nephritis is an immune complex GN that develop as a frequent complication of SLE. The pathogenesis of lupus nephritis involve a variety of pathogenic mechanisms, intra renal pathomechanisn of SLE related nephritis immune complex formation and classical complement pathway activation. Lupus nephritis doesn't develop in the absence of antinuclear antibodies. Circulating polyclonal autoantibodies bind to intrarenal nucleosomes and other autoantigen, which lead to local complement activation , cell injury and subsequent cytokine and chemokine secretion . The current management of lupus nephritis remain based on steroids, cyclophosphamide, azathioprine ,mycophenolate mefetile which are all unselective immunosuppressive drugs, these drugs have proven to be efficient in reducing lupus nephritis disease activity but the long term outcomes of lupus nephritis have not further improved during the last 30 years . Identification of renal survival is mandatory for certain purposes i.e, evaluation of efficacy of different treatment strategies among our patients and factors associated with the survival data as compared with other specialized centers.

DETAILED DESCRIPTION:
Systemic lupus erythematous is a chronic multifactorial autoimmune disease that affects many organs including kidney. Lupus nephritis is a common manifestation characterized by heterogeneous clinical and histopathological finding and often associate with poor progression and despite potent anti-inflammatory and immunosuppressive therapies still end in CKD or ESRD for too many patient. lupus nephritis is an immune complex GN that develop as a frequent complication of SLE. The pathogenesis of lupus nephritis involve a variety of pathogenic mechanisms, intra renal pathomechanisn of SLE related nephritis immune complex formation and classical complement pathway activation. Lupus nephritis doesn't develop in the absence of antinuclear antibodies. Circulating polyclonal autoantibodies bind to intrarenal nucleosomes and other autoantigen, which lead to local complement activation , cell injury and subsequent cytokine and chemokine secretion . The current management of lupus nephritis remain based on steroids, cyclophosphamide, azathioprine ,mycophenolate mefetile which are all unselective immunosuppressive drugs, these drugs have proven to be efficient in reducing lupus nephritis disease activity but the long term outcomes of lupus nephritis have not further improved during the last 30 years . Identification of renal survival is mandatory for certain purposes i.e, evaluation of efficacy of different treatment strategies among our patients and factors associated with the survival data as compared with other specialized centers.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18years old
2. Patients with SLE as defined by EULAR/ACR criteria and lupus nephritis classification according to ISN/RPS classification.
3. Available medical records for 2 and 5 years of follow up after diagnosis of lupus nephritis

Exclusion Criteria:

1. Transplant recipients
2. Pregnant females
3. Patients with combined renal pathology other than LN.
4. Those who had no baseline information in hospital medical records and had a follow up duration < 24 months will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nephrology department, Assiut University Hospital inpatient and outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of two and five years renal survival among patients with lupus nephritis | 2-5 years observation

REFERENCES:
- [Background] Mahajan A, Amelio J, Gairy K, Kaur G, Levy RA, Roth D, Bass D. Systemic lupus erythematosus, lupus nephritis and end-stage renal disease: a pragmatic review mapping disease severity and progression. Lupus. 2020 Aug;29(9):1011-1020. doi: 10.1177/0961203320932219. Epub 2020 Jun 22. PMID 32571142
- [Background] Aringer M. EULAR/ACR classification criteria for SLE. Semin Arthritis Rheum. 2019 Dec;49(3S):S14-S17. doi: 10.1016/j.semarthrit.2019.09.009. PMID 31779843
- [Background] Yu C, Li P, Dang X, Zhang X, Mao Y, Chen X. Lupus nephritis: new progress in diagnosis and treatment. J Autoimmun. 2022 Oct;132:102871. doi: 10.1016/j.jaut.2022.102871. Epub 2022 Aug 20. PMID 35999111
- [Background] Liu Y, Anders HJ. Lupus nephritis: from pathogenesis to targets for biologic treatment. Nephron Clin Pract. 2014;128(3-4):224-31. doi: 10.1159/000368581. Epub 2014 Nov 8. PMID 25401461